CLINICAL TRIAL: NCT03670524
Title: Health, Environment and Action in Louisville (HEAL) Green Heart Louisville Project
Acronym: HEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); The Nature Conservancy (Unknown)
Responsible Party: Principal Investigator, Rachel Keith, Asst Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15.1260; R01ES029846-01 (NIH)
Record Dates: First submitted 2018-08-31; First posted 2018-09-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases; Metabolic Health
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A unique pragmatic interventional trial with longitudinal follow up to assess the cardiovascular effects of increasing residential greenery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted neighborhoods for Greenness (Experimental): Using greenness as a therapeutic intervention, we will plant shrubs, grasses, young and mature trees (40-50 ft in height), so that we can evaluate changes in health and pollution, 2 years after planting.
  Interventions: Other: Greenness as a therapeutic intervention
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Greenness as a therapeutic intervention — Greenness to be used as a therapeutic intervention
  Arms: Targeted neighborhoods for Greenness

SUMMARY:
The purpose of this study is to examine how the environment and neighborhood characteristics affects the health of the area residents. The study will help determine how changing neighborhood characteristics, such as green space, affect heart health, risk factors for other diseases, sense of well- being or neighborhood cohesion.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years of age.
* Live within the targeted study location

Exclusion Criteria:

* Unwilling or unable to provide consent.
* HIV/AIDS, active treatment for cancer, active bleeding including wounds.
* Body weight less than 100 pounds or BMI>40.
* Prisoners and other vulnerable populations.
* Anyone that PI thinks is unsafe to participate in study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 835 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Analysis. Assess change from baseline arterial stiffness measurement and 2 year followup. | Baseline and 2 year followup
  Augmentation index-percent

SECONDARY OUTCOMES:
Cardiovascular Measurements. Change from Baseline Systolic and Diastolic pressures at baseline and 2 year followup. | Baseline and 2 year followup
  Blood pressure mm Hg
Physical Exam | Baseline and 2 year followup
  Body weight-pounds
Body lean mass | Baseline and 2 year followup
  Body lean mass to be measured in pounds
Body fat | Baseline and 2 year followup
  Body fat to be measured in percentage
Standing height | Baseline and 2 year followup
  standing height reported in inches
Waist, Hip measurement | Baseline and 2 year followup
  central adiposity (waist circumference, and hip circumference to be measured in inches
Respiratory status will be evaluated | Baseline and 2 year followup
  Fleisch-type pneumotachometer used to evaluate FEV1 and FVC percentages
Bucchal swab | Baseline and 2 year followup
  Assess oral microbiome and DNA from cheek swab will be stored for genetic phenotyping.
Urine collection | Baseline and 2 year followup
  metabolites of environmental volatile organic compounds ng/mg creatinine, biogenic VOCs and nicotine metabolites ng/mg creatinine, catecholamines ng/mg creatinine
Lipids | Baseline and 2 year followup
  LDL-mg/dl, HDL-mg/dl, total cholesterol-mg/dl
Toenail samples | Baseline and 2 year followup
  Toenail samples to look for heavy metal exposure
Hair samples | Baseline and 2 year followup
  Hair samples to look at cortisol levels over time.
Perceived stress scale-PSS-10 range 0-40 | Baseline and 2 year followup
  The higher the score the more perceived stress
Depression-Patient Health Questionnaire (PHQ-9) 0-27 | Baseline and 2 year followup
  The 0-4= none; 5-9= Mild, 10-14= Moderate; 15-19= moderately severe; 20-27= severe. The higher the score the more severe the depression.
Well-being assessment-Questionnaire 13-65 | Baseline and 2 year followup
  Warwick-Edinburgh Mental Well-being scale 13-65. The higher the score the higher the sense of well-being.
Health perception | Baseline and 2 year followup
  Health perception questionnaire
National Health Interview Survey tobacco questionnaire | Baseline and 2 year followup
  National Health Interview Survey tobacco questionnaire
The Alcohol Use disorders identification test (AUDIT)- Range 0-40 | Baseline and 2 year followup
  Scores of 8-15 or more are recommended indicators of hazardous and harmful alcohol use or possible alcohol dependence. Women can be lowered to a score of 7 for concern. Scores of 16-19 suggest a need for brief counseling and continues monitoring. Scores of 20 or above warrant diagnostic evaluation for alcohol dependence.
Self reported physical activity 1 | Baseline and 2 year followup
  times per week
Self reported physical activity 2 | Baseline and 2 year followup
  Exertion level of mild moderate or vigorous
Self reported education | Baseline and 2 year followup
  Education to be reported by last school grade completed
Self reported annual income | Baseline and 2 year followup
  Annual income reported by dollars
Platelet count | Baseline and 2 year followup
  cells/cubic millimeter
Complete Blood Count 1 | Baseline and 2 year followup
  White/Red blood cell count- cells per cubic millimeter
Complete Blood Count 2 | Baseline and 2 year followup
  Hemoglobin-grams/deciliter
Complete Blood Count 3 | Baseline and 2 year followup
  Hematocrit-percentage
Liver function | Baseline and 2 year followup
  AST, ALT units per liter
C-Reactive Protein | Baseline and 2 year followup
  Hs-CRP-mg/Liter

CONTACTS AND LOCATIONS:
Overall Officials: Aruni Bhatnagar, PhD, Study Director — University of Louisville; Rachel Keith, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLeish AC, Smith T, Riggs DW, Hart JL, Walker KL, Keith RJ, Anderson L, Sithu I, Pinilla-Baquero J, Srivastava S, Bhatnagar A. Community-Based Evaluation of the Associations Between Well-Being and Cardiovascular Disease Risk. J Am Heart Assoc. 2022 Nov 15;11(22):e027095. doi: 10.1161/JAHA.122.027095. Epub 2022 Nov 12. PMID 36370026